CLINICAL TRIAL: NCT01670786
Title: Safety Profile of Iodopovidone as an Agent for Pleurodesis in Malignant Pleural Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Pesquisa em Pleura e Oncologia Toracica (Network)
Collaborators: Instituto do Coracao (Other Government); Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPPOT-02
Record Dates: First submitted 2012-08-07; First posted 2012-08-22 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Pleurodesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iodopovidone 1% (Experimental): The patients enrolled in this arm were submitted to pleurodesis with iodopovidone 1% administration into pleural cavity.
  Interventions: Procedure: pleurodesis
- Iodopovidone 2% (Experimental): The patients enrolled in this arm were submitted to pleurodesis with iodopovidone 2% administration into pleural cavity.
  Interventions: Procedure: pleurodesis

INTERVENTIONS:
Procedure: pleurodesis — Comparison of two dosages of iodopovidone as an agent for pleurodesis in malignant pleural effusion

SUMMARY:
Iodopovidone is safe when using as a pleurodesis sclerosing agent for malignant pleural effusion, with minimal adverse events, especially reducing dose.

DETAILED DESCRIPTION:
Background: Chemical pleurodesis is the treatment of choice in most cases of malignant pleural effusion. The literature mentions a variety of chemicals which may be used for this purpose, each with its own advantages and disadvantages. The iodopovidone has been recently studied due to the existence of some side effects of other agents. Nevertheless, there are still some questions in the literature regarding its safety and possible adverse effects. Because of these questions, we propose the development of a study to ensure the safety and efficacy of iodopovidone as a pleurodesis sclerosing agent.

Objective: The main purpose of this study is to evaluate the safety of pleurodesis for malignant pleural effusion using iodopovidone as a sclerosing agent in different doses. The secondary objectives are to determine clinical efficacy and quality of life of the patients after realization of the proposed procedure.

Methods: There will be a randomized clinical trial, covering patients diagnosed with malignant pleural effusion at Hospital Aristides Maltez - Bahia League Against Cancer. The research was revised and approved by the Ethics in Research of the Heart Institute, Hospital das Clínicas - FMUSP and of the Hospital Aristides Maltez - Bahia League Against Cancer. The free and informed consent was evaluated by the same authority pursuant and the study group included only those who agree to participate and signed an approved. There included patients with malignant pleural effusion diagnosis. Main exclusion criteria were iodine allergia, renal failure, thyroid disease, refusal to sign the informed consent and patients unable to respond the quality of life questionnaire. After inclusion, patients were randomized and assigned to two groups according to the iodopovidone concentration solution: 1% or 2%. All procedures were performed by infusion of the solution through a chest tube previously placed.The data analysis involved clinical measures and complementary exams trying to evaluate all organ systems and sorting through possible adverse effects, classifying those as CTCAEV. Clinical measures involved MRC dyspnea schedule, analogic visual pain schedule, visual acuity test, measurement of pulse oximetry, heart rate, blood pressure and temperature. Complementary exams were chest x-ray, electrocardiogram and laboratory tests. Such measures were performed in the preoperative, immediate postoperative, second, fourth, eleventh and thirty days postoperative. Quality of life questionnaires was applied before and on thirty days postoperative as well. After that, randomized groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* malignant pleural effusion
* Recurrent pleural effusion
* Complete lung expansion (> 80%) after puncture emptying confirmed by chest radiography.
* Karnofsky index > 40.
* Agreed to participate in the study and sign an Informed Consent

Exclusion Criteria:

* Thrombocytopenia or coagulation disorders
* Patients with impaired renal function
* Pleural or active systemic infection
* Massive neoplastic infiltration of the skin
* Inability to understand the quality of life questionnaire
* Previous pleural procedures
* Allergy to iodine
* Thyroid disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety of iodopovidone as an agent for pleurodesis | Until 30th day after surgical procedure
  The safety was assessed by mean clinical measures as MRC dyspnea schedule, analogic visual pain schedule, visual acuity test, measurement of pulse oximetry, heart rate, blood pressure and temperature. Complementary exams were chest x-ray, electrocardiogram and laboratory tests.

SECONDARY OUTCOMES:
Quality of life | Until 1 week before the procedure date and 1 month after it
  Quality of life questionnaires were applied until 1 week before the procedure date and on thirty days postoperative as well.

OTHER OUTCOMES:
Efficacy of iodopovidone as an agent for pleurodesis | Procedure date and 2nd, 4th, 11st and 30th day after the surgical procedure
  The efficacy assessment was based on need of additional pleural surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M Terra, MD, PhD, Study Chair — InCor Heart Institute
Locations (1):
- Hospital Aristides Maltez, Salvador, Estado de Bahia, Brazil